CLINICAL TRIAL: NCT02086760
Title: Ultrasonography Sensibilized by Oral Hydration and Hydronephrosis in Children. Is it Useful for Diagnosis and Follow up?
Brief Title: Ultrasonography Sensibilized by Oral Hydration and Hydronephrosis in Children.
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: no subject enrolled within one year following EC and IRB approvals.
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 5580
Record Dates: First submitted 2014-02-18; First posted 2014-03-13 (Estimated); Last update posted 2015-10-02 (Estimated); Status verified 2015-10

CONDITIONS: Hydronephrosis in Children
Keywords: hydronephrosis
MeSH Terms: conditions — Hydronephrosis | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ultrasonography sensibilized by oral hydratation (Experimental): Ultrasonography before, 30 min and 90 min following hydratation.
  Interventions: Other: Ultrasonography with oral hydration; Radiation: Scintigraphy

INTERVENTIONS:
Other: Ultrasonography with oral hydration — Before, 30 min and 90 min following oral hydration
Radiation: Scintigraphy

SUMMARY:
Diagnosis and follow up of hydronephrosis is actually based on repeat ultrasonography and scintigraphy wich is a binding exam for children. We wanted to evaluate the use of ultrasonography sensibilized by an oral hydration and to determine its efficiency to detect which hydronephrosis need a surgery or not.

ELIGIBILITY:
Inclusion Criteria:

* child of 30 days old or less
* unilateral or bilateral hydronephrosis (pelvis > 5mm )

Exclusion Criteria:

* complex uropathy
* diuretic administration 6 hours prior to ultrasonography or scintigraphy
* oral feeding trouble

Max Age: 30 Days | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 0 (Actual)
Dates: Start 2014-05; Primary Completion 2016-11 (Estimated); Study Completion 2016-11 (Estimated)

PRIMARY OUTCOMES:
Similarity between the decision of the treating surgeon and the independent surgeon about the subject's medical care | V2 (Age of 6 months)
  The primary outcome measure is a composite outcome measure consisting of multiple measures.
  Indeed, the treating surgeon will make a decision (ie to operate or not) upon the clinical exam, ultrasonography with oral hydratation and scintigraphy results. The independent surgeon will only be given data from the clinical exam and the ultrasonography. For ultrasonography, the following parameters will be measured: cortical thickness, anteroposterior renal pelvis diameter, calyx diameter, kidney echogenicity, kidney size.
  The measures will be done before, 30 min and 90 min following oral hydration.
  For scintigraphy, the relative kidney function, T1/2, Tmax and NORA will be analyzed.
  The result will be reported as a single value, ie:
  * the treating surgeon's decision and the independent surgeon's decision are similar (=1) or
  * the treating surgeon's decision and the independent surgeon's decision are not similar (=0)

SECONDARY OUTCOMES:
Similarity between the decision of the treating surgeon and the independent surgeon about the subject's medical care | Between V0 (age: 30 days ) and V2 (age: 6 months)
  The secondary outcome measure is a composite outcome measure consisting of multiple measures.
  Indeed, the treating surgeon will make a decision (ie to operate or not) upon the clinical exam, ultrasonography with oral hydration and scintigraphy results. The independent surgeon will only be given data from the clinical exam and the ultrasonography with oral hydration, he will make a decision aposteriori.
  For ultrasonography, the following parameters will be measured: cortical thickness, anteroposterior renal pelvis diameter, calyx diameter, kidney echogenicity, kidney size.
  The measures will be done before, 30 min and 90 min following oral hydration.
  For scintigraphy, the relative kidney function, T1/2, Tmax and NORA will be analyzed.
  The result will be reported as a single value, ie:
  * the treating surgeon's decision and the independent surgeon's decision are similar (=1) or
  * the treating surgeon's decision and the independent surgeon's decision are not similar (=0)

CONTACTS AND LOCATIONS:
Overall Officials: Isabelle LACREUSE, MD, Principal Investigator — Hôpitaux Universitaires de Strasbourg
Locations (1):
- Service de Chirurgie Pédiatrique - Hôpital de Hautepierre- CHRU Strasbourg, Strasbourg, France